CLINICAL TRIAL: NCT01398761
Title: Development and Pilot Testing of a Web-Based, Multi-Disciplinary Sign-Out Tool to Improve Handoffs in Care
Brief Title: Development of a Sign-Out Tool to Improve Handoffs in Care
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Brigham and Women's Hospital (Other)
Collaborators: Partners Siemens Research Council (Unknown)
Responsible Party: Principal Investigator, Jeffrey L. Schnipper, MD.,MPH., Associate Professor of Medicine, Brigham and Women's Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: 2010P002915
Record Dates: First submitted 2011-07-11; First posted 2011-07-21 (Estimated); Last update posted 2014-04-28 (Estimated); Status verified 2014-04

CONDITIONS: Continuity of Patient Care; Workflow; Quality of Signout
Keywords: Continuity of patient care; Workflow; Quality of signout; Web based; Handoffs; Multi disciplinary; Written signout; Information science

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Intervention (Experimental): nurses, residents, PAs, and attendings from the two pilot services
  Interventions: Other: Signout tool

INTERVENTIONS:
Other: Signout tool — Electronic signout tool

SUMMARY:
The purpose of this grant is to fund the research necessary to fully understand the impact of this sign-out tool on clinician workflow, quality of sign-out, and continuity of care. This information will inform exactly how Partners will move ahead with tools to improve handoffs in care (i.e., whether the prototype will be adapted further, adopted Partners wide, or abandoned in favor of other solutions). The investigators hypothesize that a web-based handoff tool improves provider satisfaction, the quality of written sign-outs, and measures of continuity of care compared with current handoff tools.

DETAILED DESCRIPTION:
This study will attempt to answer the following questions:

1. What are the specific needs for clinical content among various clinical personnel (nurses, residents, and attendings) on different services at two different hospitals (MGH, BWH)?
2. How can IT support sign-out that facilitates interdisciplinary communication and yet preserves user-specific content among different clinical personnel?
3. Can a sign-out tool currently deployed at MGH be transferred to BWH using existing IT services and a minimum amount of local IS effort?
4. What will be the future needs of this tool so that it can fully access data from MetaVision once it is deployed?
5. How should the tool be further improved such that it optimizes user adoption, provider satisfaction and workflow, the quality of sign-out, and continuity of care?
6. Is it feasible for a future, refined version of this tool to be adopted across Partners acute care hospitals?

The study design is an observational, before-after pilot study. A multi-disciplinary steering committee and working group will be assembled to determine requirements and guide design in conjunction with HPM leadership, research staff, a Partners IS analyst, and MGH LCS personnel. The intervention will then be implemented on two services. Before and during implementation, several outcomes will be measured, including provider satisfaction and workflow, continuity of care, and quality of sign-out.

Deliverables will include the following:

1. Clinical and functional specifications for a new web-based sign-out tool
2. A prototype of the sign-out tool tested on 2 active clinical services, one each at MGH and BWH
3. A report of the impact of the tool on clinical care
4. Lessons learned regarding design and implementation that can be applied to more broad-based efforts
5. An update to the Sign-out White Paper with recommendations for action based on the results of this study The lessons learned will be applicable not only to Partners, but to other institutions (nationwide and worldwide) wishing to improve patient safety during handoffs in care.

ELIGIBILITY:
Inclusion Criteria:

* All nurses, residents, PAs, and attendings on the two study services

Exclusion Criteria:

* Clinical staff not on study services within study period

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 295 (Actual)
Dates: Start 2011-01; Primary Completion 2011-07 (Actual); Study Completion 2011-07 (Actual)

PRIMARY OUTCOMES:
Proportion of required data elements present | 8 months
  The proportion of required data elements present in written/typed sign-outs during tool implementation.

SECONDARY OUTCOMES:
Direct observations | 8 months
  Time spent preparing and delivering sign-out will be compared before and after implementation of the sign-out using linear regression clustered by user.
User satisfaction | 8 months
  Individual questions from the user satisfaction survey will be presented as medians with interquartile ranges on Likert-type questions and compared using the Wilcoxon rank sum test. A global satisfaction score will be derived by calculating the proportion of questions for which users were satisfied or very satisfied, and compared using linear regression. Results of the continuity of care survey will be analyzed similarly.

CONTACTS AND LOCATIONS:
Overall Officials: Jeffrey L Schnipper, MD, MPH, Principal Investigator — Brigham and Women's Hospital
Locations (1):
- Brigham & Women's Hospital, Boston, Massachusetts, United States